CLINICAL TRIAL: NCT00177294
Title: Geriatric Depression: Getting Better, Getting Well
Brief Title: Augmenting Antidepressant Treatment With Interpersonal Psychotherapy for Treating Late-life Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH037869-01 (NIH); R01MH037869 (NIH); 0404007; DATR A4-GPS
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2010-11

CONDITIONS: Depression
Keywords: Elderly; Remission; Escitalopram; Interpersonal Psychotherapy; Psychotherapy; Caregiving; Late-Life
MeSH Terms: conditions — Depression | interventions — Escitalopram; Interpersonal Psychotherapy; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants who respond partially to 6 weeks of escitalopram 10mg daily then receive 16 weeks of extension therapy with escitalopram 20 mg daily, plus weekly interpersonal psychotherapy (IPT)
  Interventions: Drug: Escitalopram; Behavioral: Interpersonal Psychotherapy
- 2 (Active Comparator): Participants who respond partially to 6 weeks of escitalopram 10mg daily then receive 16 weeks of extension therapy with escitalopram 20 mg daily, plus weekly depression care management(DCM) without interpersonal psychotherapy (IPT)
  Interventions: Drug: Escitalopram; Behavioral: Clinical Monitoring

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 mg daily for first 6 weeks, followed by escitalopram 20 mg daily for 16 additional weeks.
  Other Names: Lexapro
Behavioral: Interpersonal Psychotherapy — 16 sessions of interpersonal psychotherapy (IPT)
  Other Names: IPT
  Arms: 1
Behavioral: Clinical Monitoring — 16 weeks of depression care management(DCM). No psychotherapy will be provided.
  Arms: 2

SUMMARY:
This study will determine whether adding interpersonal psychotherapy to treatment with the antidepressant escitalopram will be more effective in reducing symptoms of depression than antidepressant medication alone.

DETAILED DESCRIPTION:
The purpose of this research study is to learn if adding psychotherapy (Interpersonal Psychotherapy) to antidepressant medication (escitalopram), will be more effective in reducing lingering symptoms of depression and decreasing the burden of these symptoms, when initial treatment with just antidepressant medication alone has led to only a partial response. Participation in the study will last up to 22 weeks.

Because fewer than 50% of elderly depressed patients achieve remission and recovery in response to first-line antidepressant pharmacotherapy, the majority of patients are left with significant symptoms and functional impairment, putting them at risk of chronic, relapsing illness, non-adherence to other medical treatment, suicide, and family caregiver burden. We will recruit and treat 320 patients with unipolar major depression aged 60 and older, using clinical management with escitalopram 10 mg/day for six weeks. Patients who are partial responders to escitalopram plus clinical management will be randomly assigned to 16 weeks of extension therapy with either 20 mg escitalopram plus clinical management or 20 mg escitalopram plus Interpersonal Psychotherapy (IPT, 16 sessions). Changes over time in measures of depressive symptoms, hopelessness, suicidal ideation, disability, and family caregiving burden will be assessed. This study will answer the question of how best to treat partial responders-by simply extending pharmacotherapy at higher doses, or by also adding psychotherapy-to remission and recovery.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00178035

http://clinicaltrials.gov/show/NCT00178074

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major depression
* Hamilton Rating Scale for Depression (HRSD) (17 item) score of 15 or higher
* Speaks English
* Willing to discontinue other psychotropic medications
* Availability of family member or other caregiver
* Hearing capacity adequate to respond to a raised conversational voice

Exclusion Criteria:

* Lifetime diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or any psychotic disorder
* Folstein Mini-Mental Status Exam (MMSE) of 17 or lower
* Suicidal
* History of treatment non-adherence in other Center protocols
* History of documented non-response to citalopram in other Center protocols
* History of non-tolerance to escitalopram therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2004-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Reynolds III, MD, Principal Investigator — University of Pittsburgh Professor of Psychiatry, Neurology, and Neuroscience
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Reynolds CF 3rd, Dew MA, Martire LM, Miller MD, Cyranowski JM, Lenze E, Whyte EM, Mulsant BH, Pollock BG, Karp JF, Gildengers A, Szanto K, Dombrovski AY, Andreescu C, Butters MA, Morse JQ, Houck PR, Bensasi S, Mazumdar S, Stack JA, Frank E. Treating depression to remission in older adults: a controlled evaluation of combined escitalopram with interpersonal psychotherapy versus escitalopram with depression care management. Int J Geriatr Psychiatry. 2010 Nov;25(11):1134-41. doi: 10.1002/gps.2443. PMID 20957693
- [Derived] Andreescu C, Tudorascu DL, Butters MA, Tamburo E, Patel M, Price J, Karp JF, Reynolds CF 3rd, Aizenstein H. Resting state functional connectivity and treatment response in late-life depression. Psychiatry Res. 2013 Dec 30;214(3):313-21. doi: 10.1016/j.pscychresns.2013.08.007. Epub 2013 Oct 18. PMID 24144505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from primary care and specialty mental-health clinics. 377 participants signed consent; 319 started study treatment; 124 were randomized. Of the 124 participants, 60 were randomized to Interpersonal Psychotherapy (IPT) and 59 randomized to Depression Care Management(DCM) without IPT.
Pre-assignment Details: 67 enrolled participants were not randomized due to the following reasons: consent withdrawal (41); did not meet eligibility criteria (16); supervening medical problems that precluded participation (4); past history of non-reponse to escitalopram (1); side effects (1).
Groups:
- Escitalopram Plus Interpersonal Psychotherapy (IPT): Participants who respond partially to 6 weeks of escitalopram 10mg daily then receive 16 weeks of extension therapy with escitalopram 20 mg daily, plus weekly interpersonal psychotherapy (IPT)
- Escitalopram Plus Depression Care Management (DCM): Participants who respond partially to 6 weeks of escitalopram 10mg daily then receive 16 weeks of extension therapy with escitalopram 20 mg daily, plus weekly depression care management without interpersonal psychotherapy (IPT)
Period: Overall Study
Arm/Group | Escitalopram Plus Interpersonal Psychotherapy (IPT) | Escitalopram Plus Depression Care Management (DCM)
Started | 60 | 64
Completed | 53 | 59
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram Plus Interpersonal Psychotherapy (IPT) | Escitalopram Plus Depression Care Management (DCM) | Total
Number analyzed (Participants) | 60 | 64 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 49 | 55 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 71.1 (7.1) | 73.4 (7.7) | 72.27 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 16 | 23 | 39
Region of Enrollment [Number; unit: participants]
  United States | 60 | 64 | 124

OUTCOME MEASURES:

1. Primary Outcome: Remission
Description: Three consecutive weekly scores of less than 7 on the Hamilton Rating Scale for Depression (N=17 item). Scores on the Hamilton Rating Scale for Depression(HRSD) range from 0 to 58, with higher scores indicating more severe depression.
Time Frame: Measured at Week 6 or 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escitalopram Plus Interpersonal Psychotherapy (IPT) | Escitalopram Plus Depression Care Management (DCM)
Number analyzed (Participants) | 60 | 64
Percentage of participants | 58 [46 to 71] | 45 [33 to 58]
Statistical Analysis 1: Comparison: Escitalopram Plus Interpersonal Psychotherapy (IPT) vs Escitalopram Plus Depression Care Management (DCM); We conducted Cox regreassion analyses of time to remission and logistic modeling for rates of remission. We tested group difference in Hamilton depession ratings over time via mixed-effects modeling; Test type: Superiority or Other; p = 0.14, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Escitalopram Plus Interpersonal Psychotherapy (IPT) | Escitalopram Plus Depression Care Management (DCM)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/64
Other Adverse Events (participants affected / at risk) | 0/60 | 0/64

LIMITATIONS AND CAVEATS:
The study design does not allow an inference about which specific intervention led to further improvement. Was it simply a dose increase of escitalopram from 10mg to 20mg? Is this intensive contact necessary for improvement?

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No